CLINICAL TRIAL: NCT03288883
Title: Fractional Microablative CO2-laser Versus Photothermal Non-ablative Erbium:YAG-laser for the Management of Genitourinary Syndrome of Menopause: A Non-inferiority, Single-blind Randomised Controlled Trial
Brief Title: RCT of Laser Therapy for GSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCTGSM
Record Dates: First submitted 2017-09-07; First posted 2017-09-20 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fractional Microablative CO2-laser (Active Comparator)
  Interventions: Device: Fractional Microablative CO2-laser
- Photothermal Non-ablative Erbium:YAG-laser (Active Comparator)
  Interventions: Device: Photothermal Non-ablative Erbium:YAG-laser

INTERVENTIONS:
Device: Photothermal Non-ablative Erbium:YAG-laser — Laser treatment of the vagina for GSM
  Arms: Photothermal Non-ablative Erbium:YAG-laser
Device: Fractional Microablative CO2-laser — Laser treatment of the vagina for GSM
  Arms: Fractional Microablative CO2-laser

SUMMARY:
The aim of the current study is to assess whether the CO2-laser results in superior alleviation of GSM symptoms compare to Er:YAG-laser. Specifically, we will compare objective and subjective measurements of symptoms and clinical signs of GSM, between groups of postmenopausal women with GSM receiving treatment with CO2-laser or Er:YAG-laser.

DETAILED DESCRIPTION:
Genitourinary Syndrome of Menopause (GSM) is the new terminology for "vulvovaginal (VVA)". Although women may present with some or all of the clinical signs and symptoms, the most common symptom of VVA/GSM is vaginal dryness. Vaginal dryness appears early at menopause with a subsequent increase of prevalence as postmenopausal years' progresses and is associated with rising occurrence of lower urinary tract symptoms (LUTS).

The therapeutic management of GSM includes lubricants and moisturizers as a first line therapy and low-dose vaginal estrogens as a second one, especially for women with a history of estrogen dependent cancer. However, lubricants and moisturizers can only be used for symptoms relief during sexual intercourse. They do not restore the local pathophysiology and they are inefficacious when LUTS are present. However, the quality of evidence is low or very-low when estrogens efficacy is compared to placebo, while the risk to the endometrial thickness with sustained vaginal estrogen use is not clear.

Recently, intravaginal laser therapy has been proposed for the management of GSM. There are currently two lasers available. All available studies consistently suggest that both lasers (CO2-laser and Er:YAG-laser) are safe and have a high efficacy on alleviating vaginal dryness and dyspareunia, as well as restoring the local pathophysiology. Additionally, data regarding CO2-laser indicate LUTS improvement, as well as sexual function-satisfaction and quality of women's life. Relevant published data are not available for the Er:YAG-laser. Moreover, there is lack of studies comparing the 2 laser-technologies for the management of postmenopausal women with GSM.

The aim of the current study is to assess whether the CO2-laser results in superior alleviation of GSM symptoms compare to Er:YAG-laser. Specifically, we will compare objective and subjective measurements of symptoms and clinical signs of GSM, between groups of postmenopausal women with GSM receiving treatment with CO2-laser or Er:YAG-laser.

ELIGIBILITY:
Inclusion Criteria:

1. Dryness and dyspareunia with moderate to severe intensity
2. Vaginal Health Index <15
3. Absence of menstruation for at least 12 months
4. Recent Negative Pap-smear test (For women over 65 years old a negative pap smear test up to the age of 65).

Exclusion Criteria:

1. Not willing to abstain from vaginal intercourse for one week following the laser-therapy
2. Use of hormonal therapy within 6 months prior to study inclusion (systemic or local)
3. Acute urinary tract infections (UTIs)
4. History of a genital fistula, a thin recto-vaginal septum as determined by the investigator or history of a fourth-degree laceration during screening physical exam (e.g., perineal body)
5. Active sexually transmitted disease upon vaginal exam (as determined by the investigator) that precludes treatment or any other vaginal infection
6. Active or history of genital herpes
7. Prolapse stages > II (according to the POP-Q system)
8. History of radiotherapy for cervical or uterine cancer
9. Medical condition that may interfere with participants' compliance to the protocol

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Dryness - 10cm visual analogue scale | 1 year
Dyspareunia- 10cm visual analogue scale | 1 year
Itching- 10cm visual analogue scale | 1 year
Burning- 10cm visual analogue scale | 1 year
Dysuria- 10cm visual analogue scale | 1 year
Frequency- 10cm visual analogue scale, | 1 year
Urgency-10cm visual analogue scale | 1 year
Urinary incontinence- 10cm visual analogue scale | 1 year
Overall sexual satisfaction- Female sexual function index | 1 year
Frequency- 3 day voiding diary | 1 year
Urgency- 3 day voiding diary, | 1 year
Urinary incontinence- 3 day voiding diary | 1 year
Overall sexual satisfaction- 10cm visual analogue scale | 1 year
Overall sexual satisfaction- frequency of sexual intercourse, | 1 year

SECONDARY OUTCOMES:
Quality of life- patients global impression of improvement questionnaire | 1 year
Quality of life- day to day impact of vaginal ageing questionnaire | 1 year
Quality of life- kings health questionnaire | 1 year
Global impression of improvement- day to day impact of vaginal ageing questionnaire | 1 year
Global impression of improvement- patients global impression of improvement questionnaire | 1 year
Global impression of improvement- kings health questionnaire | 1 year
Vaginal health index score- 5 components, elasticity, epithelial integrity, pH, moisture and fluid volume | 1 year
Vaginal maturation value- vaginal smear stained with papanicolaou technique and VMI value is evaluated by defining the percentage of superficial, intermediate and paranasal epithelial cells on smear. | 1 year
  VMV = ((1x%superficial)+(0.5x%intermediate)+0xparabasal))

CONTACTS AND LOCATIONS:
Locations (1):
- Urogynaecology Department, King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No